CLINICAL TRIAL: NCT05468060
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics of Single Ascending Dose (SAD) of PA1010 Tablets in Chinese Healthy Subjects and the Effects of Food and Gender on Pharmacokinetics
Brief Title: Study of the Safety, Tolerability, Pharmacokinetic Characteristics of PA1010 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Palo Alto Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PA1010-101
Record Dates: First submitted 2022-07-12; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Chronic HBV Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- PA1010 5mg (Experimental): Ten subjects will be randomly assigned in a ratio of 4:1 to receive 5 mg of PA1010 tablets or 5mg of PA1010 placebo tablets. They will be administered a single dose and observed for four days.
  Interventions: Drug: PA1010
- PA1010 10mg (Experimental): Ten subjects will be randomly assigned in a ratio of 4:1 to receive 10mg of PA1010 tablets or 10mg of PA1010 placebo tablets. They will be administered a single dose and observed for four days.
  Interventions: Drug: PA1010
- PA1010 20mg (Experimental): Ten subjects will be randomly assigned in a ratio of 4:1 to receive 20mg of PA1010 tablets or 20mg of PA1010 placebo tablets. They will be administered a single dose and observed for four days.
  Interventions: Drug: PA1010
- PA1010 30mg (Experimental): Ten subjects will be randomly assigned in a ratio of 4:1 to receive 30mg of PA1010 tablets or 30mg of PA1010 placebo tablets. They will be administered a single dose and observed for four days.
  Interventions: Drug: PA1010
- PA1010 45mg (Experimental): Ten subjects will be randomly assigned in a ratio of 4:1 to receive 45mg of PA1010 tablets or 45mg of PA1010 placebo tablets. They will be administered a single dose and observed for four days.
  Interventions: Drug: PA1010
- PA1010 60mg (Experimental): Ten subjects will be randomly assigned in a ratio of 4:1 to receive 60mg of PA1010 tablets or 60mg of PA1010 placebo tablets. They will be administered a single dose and observed for four days.
  Interventions: Drug: PA1010
- PA1010 10mg before and after meals (Experimental): Ten subjects will be administered 10mg PA1010 after overnight fasting for 10 hours in the first cycle, and then will be administered 10mg PA1010 within 30 minutes after high-fat meal in the second cycle. They will receive a single dose in each cycle and will be observed for four days. The cleaning period between the two cycles is 10 days.
  Interventions: Drug: PA1010
- PA1010 10mg after and before meals (Experimental): Ten subjects will be administered 10mg PA1010 within 30 minutes after the high-fat meal in the first cycle, and then will be administered 10mg PA1010 after overnight fasting 10 hours in the second cycle. They will receive a single dose in each cycle and will be observed for four days. The cleaning period between the two cycles is 10 days.
  Interventions: Drug: PA1010

INTERVENTIONS:
Drug: PA1010 — Placebo as control

SUMMARY:
The primary objectives of this study are to evaluate the safety, tolerability and pharmacokinetics characteristics of single ascending dose (SAD) of PA1010 tablets in Chinese healthy adults and the impact of food and gender on the pharmacokinetics

DETAILED DESCRIPTION:
Stage I: Single dose, Single Ascending Dose (SAD)

This is a randomized, double-blind, placebo-controlled, dose-escalation clinical trial. The objective is to evaluate the safety, tolerability and pharmacokinetics characteristics of PA1010 tablets in Chinese healthy subjects. There are six dose groups of PA1010 ( 5 mg、10 mg、20 mg、30 mg、45 mg and 60 mg) proposed to be tested sequentially in this study. A total of 60 healthy subjects are planned to be enrolled in this study and will be randomly assigned to the corresponding dose group in equal proportion, stratified by gender (male vs female). 10 subjects in each dose group are randomly assigned in a ratio of 4:1 to receive PA1010 tablets or placebo. All subjects will be dosed in a single dose, and the dose-related safety, tolerability and PK of PA1010 will be evaluated.

Stage II: Study on the effect of food on Pharmacokinetics

This is a single center, randomized, open, two group crossover, self-control clinical trial. A total of 20 subjects are planned to be enrolled in this study, and will be randomly assigned to a dosing order (i.e. fasting administration followed by high-fat meal administration, or high-fat meal administration followed by fasting administration) in a ratio of 1:1. Subjects will be dosed 10 mg PA1010 tablets in a single dose, and the food-related PK of PA1010 will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged between 18 and 55 (including upper and lower limits);
2. Body mass index (BMI) is between 18 and 28 kg/m2 (including upper and lower limits);
3. During the study period (from signing the informed consent to the last follow-up) and within 90 days after the last dose, there is no possibility of pregnancy (or making the sexual partner pregnant), childbirth or lactation, including:

   1. Menopausal women who have menopause for more than 12 months or undergo sterilization (such as hysterectomy or bilateral ovariectomy);
   2. Postmenopausal women, who have negative urine pregnancy test within 24 hours before the first dose, are willing to take more than one effective contraceptive method from the screening period to 90 days after the last dose, including intrauterine device, fallopian tube ligation, double barrier method (condom / vaginal diaphragm + spermicide) and male partner vas deferens ligation, but do not include oral contraceptives;
   3. Men are willing to take more than one effective contraceptive method from the first dose to 90 days after the last dose, including vasectomy, double barrier method, female partner's use of contraceptives, intrauterine device or tubal ligation, etc.;
   4. Avoid sex during the study period to 90 days after the last dose;
4. There is no history of major diseases, and the physical examination, vital signs, electrocardiogram and laboratory examination results during the screening period are normal, or although they exceed the normal reference value range, they are judged by the researcher to be of no clinical significance;
5. Be able to communicate with clinical staff normally and comply with the requirements of this study;
6. Sign the informed consent form to indicate willingness to participate in this study.

Exclusion Criteria:

1. Any medical condition that the investigator considers to be likely to increase the risk of study participation (in particular, a history of esophageal or gastrointestinal ulcers), that may interfere with drug absorption, distribution, metabolism, or excretion, or that may impair adherence to the study protocol;
2. Those who have received any other study drug within 90 days before the first dose of the study drug;
3. Those who have received other prescription or over-the-counter drugs that will effect the study evaluation considered by the investigator that within 14 days prior to the first administration of the study drug (or within 5 half-lives of the drug, whichever is longer）；
4. Those who have donated blood or lost a lot of blood (>400 ml) within 3 months before the first dose of the study drug;
5. Major surgery or great trauma within 6 months before the first dose of the study drug (the investigator make the judgement based on the previous medical history);
6. Consumption of beverages or foods containing grapefruit, pomegranate, papaya, grapes, carambola within 14 days, or do not agree to refrain from taking those beverages or foods every day during the study；
7. Any alcoholic products within 48 hours before the first administration of the study drug, or disagree to refrain from taking any alcohol products every day during the study;
8. Any foods or beverages rich in caffeine and xanthine within 48 hours before the first dose of the study drug(coffee, tea, coke, chocolate, seafood, animal liver, etc.) or disagree to refrain from taking those foods and beverages every day during the study;
9. Abnormal ECG during screening or baseline period, which is judged to be clinically significant by the investigator; Or QTcF > 450 ms during screening or baseline period；
10. History of heart disease, including a family history of sudden death caused by cardiac causes or QT interval prolongation syndrome;
11. History of serious kidney disease (judged by the investigator);
12. Difficulty in venous blood collection, or known to have a history of needle fainting and blood fainting for many times;
13. Clinical or laboratory evidence shows that there is one of the following situations: hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV), syphilis carrying / infection;
14. Any history of food and drug allergy of clinical significance judged by the investigator;
15. Any history of drug abuse or urine drug test (+) in the screening period within 1 year before the first administration of the study drug;
16. Regular drinking history within 6 months before screening. Women have more than 7 cups / week, men have more than 14 cups / week (1 cup =5 ounces of wine or 12 ounces of beer or 1.5 ounces of spirits) or the alcohol test exceeds the standard during the screening period;
17. Those who cannot quit smoking as required during the study period or whose cigarette test paper (urine nicotine test) is positive during the screening period;
18. Participated in this study before.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-06-28 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects having abnormal hematology laboratory parameters | Up to 72 hours after last dose
  Absolute and relative number of subjects with values below, within or above the normal range will be assessed.
Number of subjects with abnormal clinical chemistry parameters | Up to 72 hours after last dose
  Absolute and relative number of subjects with values below, within or above the normal range will be assessed.
Number of subjects with abnormal values for urinalysis | Up to 72 hours after last dose
  Absolute and relative number of subjects with values below, within or above the normal range will be assessed.
Number of subjects with abnormal with blood coagulation function | Up to 72 hours after last dose
  Absolute and relative number of subjects with values below, within or above the normal range will be assessed.
Ear temperature | Up to 72 hours after last dose
  Vital sign-ear temperature
Systolic and diastolic blood pressure | Up to 72 hours after last dose
  Vital sign-Systolic and diastolic blood pressure
Pulse rate | Up to 72 hours after last dose
  Vital sign-Pulse rate
Breathing rate | Up to 72 hours after last dose
  Vital sign-Breathing rate
ECG parameter-QTc interval | Up to 72 hours after last dose
  A 12 lead electrocardiogram (ECG) will be recorded using an ECG machine that automatically calculates the QTc intervals
ECG parameter-PR interval | Up to 72 hours after last dose
  A 12 lead electrocardiogram (ECG) will be recorded using an ECG machine that automatically measures PR intervals
ECG parameter-QRS duration | Up to 72 hours after last dose
  A 12 lead electrocardiogram (ECG) will be recorded using an ECG machine that automatically measures QRS duration
Number of subjects experiencing adverse events (AEs) | Up to 4days after the last dose
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical study subject administered a medicinal product which does not necessarily have a causal relationship with this treatment.
Pharmacokinetics of single dose of PA1010-Cmax | Up to 72 hours after last dose
  Blood samples will be collected serially, and the concentrations of PA1010 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Maximum Observed Plasma Concentration (Cmax)
Pharmacokinetics of single dose of PA1010-Tmax | Up to 72 hours after last dose
  Blood samples will be collected serially, and the concentrations of PA1010 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Time to Reach Maximum Observed Plasma Concentration (Tmax)
Pharmacokinetics of single dose of PA1010-AUC | Up to 72 hours after last dose
  Blood samples will be collected serially, and the concentrations of PA1010 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Area Under the Plasma Concentration-Time Curve (AUC)

SECONDARY OUTCOMES:
Pharmacokinetics of single dose of PA1010-T1/2 | Up to 72 hours after last dose
  Blood samples will be collected serially, and the concentrations of PA1010 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Elimination Half-Life Period (T1/2）
Pharmacokinetics of single dose of PA1010-Vz/F | Up to 72 hours after last dose
  Blood samples will be collected serially, and the concentrations of PA1010 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Apparent Volume of Distribution(Vz/F)
Pharmacokinetics of single dose of PA1010-λz | Up to 72 hours after last dose
  Blood samples will be collected serially, and the concentrations of PA1010 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Elimination Rate Constant(λz)
Pharmacokinetics of single dose of PA1010-CL/F | Up to 72 hours after last dose
  Blood samples will be collected serially, and the concentrations of PA1010 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Apparent Clearance(CL/F)

CONTACTS AND LOCATIONS:
Overall Officials: Xuebing Yan, MD, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China